CLINICAL TRIAL: NCT06018025
Title: New Daily Persistent Headache (NDPH): Biomarker Study and Therapy in Children and Adolescents
Brief Title: NDPH Biomarker Study in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: International Headache Society (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00113907
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: New Persistent Daily Headache
Keywords: NPDH; CGRP; PACAP; BDNF; NGF; TNF-alpha; VIP; biomarker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Biospecimen Retention: Samples Without DNA — whole blood, serum,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NPDH (New Persistent Daily Headache): Patients with new persistent daily headache (NDPH) ages 10-18 years will be recruited and consented by the study coordinator. Patients will be recruited from patients already established with the Duke Pediatric Neurology clinic with a diagnosis of NDPH, or after their initial visit to establish the diagnosis of NDPH through the Duke, pediatric neurology clinics, personal communication and networking, and through the Duke adult headache clinic.
  Interventions: Drug: CGRP antibody
- Healthy (Normal) Controls: Children with normal development, aged 10-18 years, will be identified via the electronic health records of well-child visits in Duke Children's Hospital, community advertising and through networking with colleagues and friends.
  Exclusion: 1) History of concussion or head injury 2) Psychiatric disorders 3) History of migraines or other headache disorder treated in the past 4) Known structural brain lesions (tumor, hydrocephalus, congenital anomalies)
- Chronic Migraine: Patients between 10-18 yrs of age:
  A) Headache (migraine-like or tension-type-like) on ≥15 days/month for >3 months, and fulfilling criteria B and C, B) Occurring in a patient who has had at least five attacks fulfilling criteria B-D for 1.1 Migraine without aura and/or criteria B and C for 1.2 Migraine with aura C) On ≥8 days/month for >3 months, fulfilling any of the following (1) criteria C and D for 1.1 Migraine without aura 2) criteria B and C for 1.2 Migraine with aura 3) believed by the patient to be migraine at onset and relieved by a triptan or ergot derivative D) Not better accounted for by another ICHD-3 diagnosis
  Interventions: Drug: CGRP antibody

INTERVENTIONS:
Drug: CGRP antibody — treatment with CGRP antibody for 4 months
  Groups: Chronic Migraine; NPDH (New Persistent Daily Headache)

SUMMARY:
This study will recruit pediatric patients with NDPH (New Daily Persistent Headache), characterize their headache in a standard manner, and treat the NDPH with standard medications used for treatment of headaches in this population. Response to treatment with CGRP blocking Ab medications will be evaluated. Biomarkers related to headache disorders will be measured before and after treatment.

DETAILED DESCRIPTION:
Subjects age 10-18 with diagnosis of NDPH (International Classification of Headache Disorders D ICHD-3 criteria) will be recruited for the study. Consenting subjects will receive standard headache care and treatment, including treatment with CGRP Blocking Ab medications. Blood will be drawn before and after treatment, with assessment of Calcitonin Gene Related Peptid, Pituitary Adenylate Cyclase Activating Peptid (PACAP), Brain derived Neurotrophic factor (BDNF), Nerve Growth Factor (NGF), and Tumor Necrosis Factor alpha, and Vasointestinal peptic (VIP) before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 10-18 yo with diagnosis of new daily persistent headache (ICHD-3 criteria) who have normal developmental history for age
* Subject and parent legal guardian able to communicate in English, understand and consent to study
* Subject will to undergo monthly injections at home for treatment of NDPH
* Normal neuro imaging
* No prior treatment with CGRP blocking medications or botulinum toxin

Exclusion Criteria:

* History of Reynauds syndrome
* History of concussion or prior neurosurgery
* Any structural brain lesion including hydrocephalus, congenital anomalies (including chiari malformation)
* History of psychiatric disorders
* History of any headache disorder (including migraine) prior to the diagnosis of NDPH
* Pregnancy
* Prior treatment with any CGRP blocking medication
* Treatment with Botulinum toxin injections previously
* Any other condition that in the opinion of the PI would interfere with the planned study treatment

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 10 patients with NPDH age 10-18yrs 10 patients with chronic migraine age 10-18 yrs 10 normal controls age 10-18 yrs
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Change in Calcitonin Gene Related Peptide (CGRP) levels in blood | baseline and 4 months
  biomarker
Change in Pituitary Adenylate Cyclase-activating Peptide (PACAP) levels in blood | baseline and 4 months
  protein biomarker
Change in Brain derived Neurotrophic factor (BDNF) levels in blood | baseline and 4 months
  protein biomarker
Change in Nerve Growth Factor (NGF) levels in blood | baseline and 4 months
  protein biomarker
Change in Tumor Necrosis Factor alpha levels in blood | baseline and 4 months
  protein biomarker
Change in Vaso Intestinal peptide(VIP) levels in blood | baseline and 4 months
  protein biomarker

SECONDARY OUTCOMES:
Disability Scoring | 0 to 4 months
  Changes in the Disability Scoring using the Pediatric Migraine Disability Assessment(PedMIDAS) will be recorded at the baseline visit (prior to first CGRP-AB treatment) and 4 months after receiving CGRP-AB treatment. Disability Grade ; 0 to 10. Little to none ; 11 to 30. Mild ; 31 to 50. Moderate ; Greater than 50. Severe
Change in Headache frequency | 0 to 4 months
  Self-reported headache frequency will be recorded as the number of headaches in the prior month, collected at baseline and 4 months after last CGRP-AB treatment. The patients will be encouraged to keep a headache diary.
Screen for Child Anxiety Related Disorders (SCARED) | at enrollment
  41 items and 5 factors that parallel the DSM-IV classification of anxiety disorders. A total score of 0-9, normal or no anxiety; 10-18, mild to moderate anxiety; 19-29, moderate to severe anxiety; and 30-63, severe anxiety.
Patient Health Questionnaire-9 modified for Adolescents administered after recruitment | at enrollment
  Scores of 0-4 points normal or minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression and 20-27 severe depression
Change in Headache Pain Intensity | 0 to 4 months
  Average severity will be measured using a 10-point pain scale, where a higher score indicates greater pain.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Werner, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greene KA, Gentile CP, Szperka CL, Yonker M, Gelfand AA, Grimes B, Irwin SL. Calcitonin Gene-Related Peptide Monoclonal Antibody Use for the Preventive Treatment of Refractory Headache Disorders in Adolescents. Pediatr Neurol. 2021 Jan;114:62-67. doi: 10.1016/j.pediatrneurol.2020.09.014. Epub 2020 Oct 5. PMID 33232919
- [Background] Demartini C, Francavilla M, Zanaboni AM, Facchetti S, De Icco R, Martinelli D, Allena M, Greco R, Tassorelli C. Biomarkers of Migraine: An Integrated Evaluation of Preclinical and Clinical Findings. Int J Mol Sci. 2023 Mar 10;24(6):5334. doi: 10.3390/ijms24065334. PMID 36982428
- [Background] Gelfand AA, Robbins MS, Szperka CL. New Daily Persistent Headache-A Start With an Uncertain End. JAMA Neurol. 2022 Aug 1;79(8):733-734. doi: 10.1001/jamaneurol.2022.1727. No abstract available. PMID 35788252
- [Background] Goadsby PJ. New daily persistent headache: a syndrome, not a discrete disorder. Headache. 2011 Apr;51(4):650-3. doi: 10.1111/j.1526-4610.2011.01872.x. PMID 21457252
- [Background] Peng KP, Rozen TD. Update in the understanding of new daily persistent headache. Cephalalgia. 2023 Feb;43(2):3331024221146314. doi: 10.1177/03331024221146314. PMID 36759317
- [Background] Gladstein J, Holden EW. Chronic daily headache in children and adolescents: a 2-year prospective study. Headache. 1996 Jun;36(6):349-51. doi: 10.1046/j.1526-4610.1996.3606349.x. PMID 8707551
- [Background] Hanci F, Kilinc YB, Kilinc E, Turay S, Dilek M, Kabakus N. Plasma levels of vasoactive neuropeptides in pediatric patients with migraine during attack and attack-free periods. Cephalalgia. 2021 Feb;41(2):166-175. doi: 10.1177/0333102420957588. Epub 2020 Sep 9. PMID 32903061
- [Background] Evers S. CGRP in Childhood and Adolescence Migraine: (Patho)physiological and Clinical Aspects. Curr Pain Headache Rep. 2022 Jun;26(6):475-480. doi: 10.1007/s11916-022-01047-5. Epub 2022 Mar 30. PMID 35353359
- [Background] Christensen CE, Ashina M, Amin FM. Calcitonin Gene-Related Peptide (CGRP) and Pituitary Adenylate Cyclase-Activating Polypeptide (PACAP) in Migraine Pathogenesis. Pharmaceuticals (Basel). 2022 Sep 27;15(10):1189. doi: 10.3390/ph15101189. PMID 36297301
- [Background] Vollesen ALH, Amin FM, Ashina M. Targeted Pituitary Adenylate Cyclase-Activating Peptide Therapies for Migraine. Neurotherapeutics. 2018 Apr;15(2):371-376. doi: 10.1007/s13311-017-0596-x. PMID 29464574
- [Background] Sarchielli P, Caproni S, Costa C, Szok D, Tajti J. Chapter 10: Biochemistry of Primary Headaches. Pathophysiology of Headaches 2015: 185-216.
- [Background] Ashina M, Terwindt GM, Al-Karagholi MA, de Boer I, Lee MJ, Hay DL, Schulte LH, Hadjikhani N, Sinclair AJ, Ashina H, Schwedt TJ, Goadsby PJ. Migraine: disease characterisation, biomarkers, and precision medicine. Lancet. 2021 Apr 17;397(10283):1496-1504. doi: 10.1016/S0140-6736(20)32162-0. Epub 2021 Mar 25. PMID 33773610
- [Background] Moyes C, Belaghi R, Webster RJ, Whitley N, Pohl D. Cognitive Behavioral Therapy for Children With Headaches: Will an App Do the Trick? J Child Neurol. 2023 Mar;38(3-4):169-177. doi: 10.1177/08830738231170067. Epub 2023 Apr 25. PMID 37097885
- [Background] McAbee GN, Morse AM, Assadi M. Pediatric Aspects of Headache Classification in the International Classification of Headache Disorders-3 (ICHD-3 beta version). Curr Pain Headache Rep. 2016 Jan;20(1):7. doi: 10.1007/s11916-015-0537-5. PMID 26749046
- [Background] Begasse de Dhaem O, Rizzoli P. Refractory Headaches. Semin Neurol. 2022 Aug;42(4):512-522. doi: 10.1055/s-0042-1757925. Epub 2022 Nov 2. PMID 36323303
- [Background] Nierenburg H, Newman LC. Update on New Daily Persistent Headache. Curr Treat Options Neurol. 2016 Jun;18(6):25. doi: 10.1007/s11940-016-0408-3. PMID 27080086
- [Background] Mack KJ. What incites new daily persistent headache in children? Pediatr Neurol. 2004 Aug;31(2):122-5. doi: 10.1016/j.pediatrneurol.2004.02.006. PMID 15301832
- [Background] Li D, Rozen TD. The clinical characteristics of new daily persistent headache. Cephalalgia. 2002 Feb;22(1):66-9. doi: 10.1046/j.1468-2982.2002.00326.x. PMID 11993616
- [Background] Baron EP, Rothner AD. New daily persistent headache in children and adolescents. Curr Neurol Neurosci Rep. 2010 Mar;10(2):127-32. doi: 10.1007/s11910-010-0097-3. PMID 20425237
- [Background] Mozafarihashjin M, Togha M, Ghorbani Z, Farbod A, Rafiee P, Martami F. Assessment of peripheral biomarkers potentially involved in episodic and chronic migraine: a case-control study with a focus on NGF, BDNF, VEGF, and PGE2. J Headache Pain. 2022 Jan 6;23(1):3. doi: 10.1186/s10194-021-01377-6. PMID 34991456